CLINICAL TRIAL: NCT03479463
Title: A Matched Case Clinical Registry - Efficacy of AmnioFix in the Prevention of Post-Operative Salivary Leaks Following Head and Neck Surgery
Brief Title: Use of Human Dehydrated Amnion Chorion Allograft in Laryngectomy/Pharyngectomy
Status: Terminated | Type: Observational
Why Stopped: Slow enrollment
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AFSUR003
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Larynx Cancer; Pharynx Cancer; Pharyngocutaneous Fistula
MeSH Terms: conditions — Laryngeal Neoplasms; Pharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 150 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment with Dehydrated Human Amnion Chorion Allograft
  Interventions: Biological: Dehydrated human amnion/chorion membrane
- Standard of Care

INTERVENTIONS:
Biological: Dehydrated human amnion/chorion membrane — Laryngectomy/pharyngectomy patched with dehydrated human amnion chorion allograft
  Groups: Treatment with Dehydrated Human Amnion Chorion Allograft

SUMMARY:
This trial aims to determine if intra-operative use of human dehydrated amnion chorion allograft improves post-operative patient healing outcomes.

DETAILED DESCRIPTION:
This study is to determine if intra-operative use of Amnio-Fix improves post-operative patient healing outcomes after laryngectomy and/or pharyngectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is scheduled to undergo laryngectomy and/or pharyngectomy procedure due to oncological indication
2. Subject is age 18 or older
3. Subject is willing and able to provide informed consent and participate in all procedures and follow-up evaluations necessary to complete the study

Exclusion Criteria:

1. Subjects currently enrolled in or planning to enroll in another clinical trial
2. Subjects with a known history of poor compliance with medical treatments
3. Subjects that are using or have used an investigational drug, device, or biologic within the 12 weeks prior to treatment
4. Subjects that have any significant medical condition(s) that, in the opinion of the Investigator, would interfere with protocol evaluation and participation
5. Subject has undergone previous pharyngeal reconstructive surgery
6. Pregnancy at enrollment or within last 6 months, women who are breastfeeding, or women of childbearing potential who are planning to become pregnant during the time of the study OR are unwilling/unable to use acceptable methods of contraception (birth control pills, barriers, or abstinence)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a single-center, matched case registry. The medical records of approximately 40 patients meeting all documentation and eligibility requirements will comprise the retrospective cohort. A total of 40 subjects will be enrolled prospectively at Mount Sinai Hospital. It is expected that the majority of the subjects will be recruited through the investigators' standard admission practices. All subjects selected for the study will not be excluded because of race or ethnicity and all efforts will be made to adequately represent the patient population in the area in which they are chosen.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Pharayngocutaneous Fistula Development (PCF) | 60 days
  Incidence of PCF developement necessitating intervention within the 60 day time point.

CONTACTS AND LOCATIONS:
Overall Officials: Brett Miles, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, New York, New York, United States